CLINICAL TRIAL: NCT02000583
Title: Effect of Aerobic Exercise on Pathophysiology of PreClinical Alzheimer's Disease
Brief Title: Alzheimer's Prevention Through Exercise
Acronym: APEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13376; R01AG043962-01 (NIH)
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; AD; Aerobic Exercise; Exercise
MeSH Terms: conditions — Alzheimer Disease; Motor Activity | interventions — Exercise; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise Group (Experimental): Exercise 150 minutes per week (over 3 to 5 days) for 52 weeks
  Interventions: Other: Aerobic Exercise
- Control Group (Other): Standard of Care exercise recommendations
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Aerobic Exercise — Aerobic group participants will engage in 150 minutes of aerobic exercise over 4-5 days per week for 52 weeks
  Arms: Aerobic Exercise Group
Other: Standard of Care — Control group participants will be provided educational materials on starting an exercise program, but will receive no formal support for their exercise program.
  Other Names: Standard of Care for exercise recommendations
  Arms: Control Group

SUMMARY:
The purpose of this study is to learn about the possible benefits of aerobic exercise in controlling or reducing the amount of amyloid present in the brain, reducing changes in brain structure that may lead to Alzheimer's Disease (AD), and increasing cognitive ability in individuals that have amyloid deposits and are at risk to develop AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Dementia Rating 0 (nondemented)
* Age 65 or older
* Florbetapir PET evidence of cerebral amyloidosis
* Sedentary or underactive by the Telephone Assessment of Physical Activity
* Stable doses of medications for 30 days.
* Clinician judgment regarding subject's health status and likelihood to successfully complete the 1-year exercise intervention

Exclusion Criteria:

* Clinically significant major psychiatric disorder (e.g., Major Depressive Disorder) according to standard criteria or significant psychiatric symptoms that could impair the completion of the study
* Clinically-significant systemic illness that may affect safety or completion of the study
* History of clinically-evident stroke
* Clinically-significant infection within the last 30 days
* Active cardiac condition (e.g. angina, myocardial infarction, atrial fibrillation) or pulmonary condition in the past 2 years that, in the investigator's opinion, could pose a safety risk to the participant-unless cleared for exercise by the participant's primary care physician or cardiologist.
* Uncontrolled hypertension within the last 6 months
* History of cancer in the last 5 years (except non-metastatic basal or squamous cell carcinoma)
* History of drug or alcohol abuse as defined by DSM-IV criteria within the last 2 years
* Insulin-dependent diabetes mellitus
* Significant pain or musculoskeletal disorder prohibiting participation in an exercise program
* Unwillingness to undergo or contraindication to brain MRI scan.
* History within the last 5 years of primary or recurrent malignant disease with the exception of resected localized cutaneous squamous cell carcinoma, basal cell carcinoma, cervical carcinoma, or prostate cancer.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-11; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Burns, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Taylor MK, Sullivan DK, Morris JK, Vidoni ED, Honea RA, Mahnken JD, Burns JM. High Glycemic Diet Is Related to Brain Amyloid Accumulation Over One Year in Preclinical Alzheimer's Disease. Front Nutr. 2021 Sep 27;8:741534. doi: 10.3389/fnut.2021.741534. eCollection 2021. PMID 34646853
- [Derived] Kaufman CS, Honea RA, Pleen J, Lepping RJ, Watts A, Morris JK, Billinger SA, Burns JM, Vidoni ED. Aerobic exercise improves hippocampal blood flow for hypertensive Apolipoprotein E4 carriers. J Cereb Blood Flow Metab. 2021 Aug;41(8):2026-2037. doi: 10.1177/0271678X21990342. Epub 2021 Jan 28. PMID 33509035
- [Derived] Vidoni ED, Morris JK, Watts A, Perry M, Clutton J, Van Sciver A, Kamat AS, Mahnken J, Hunt SL, Townley R, Honea R, Shaw AR, Johnson DK, Vacek J, Burns JM. Effect of aerobic exercise on amyloid accumulation in preclinical Alzheimer's: A 1-year randomized controlled trial. PLoS One. 2021 Jan 14;16(1):e0244893. doi: 10.1371/journal.pone.0244893. eCollection 2021. PMID 33444359
- [Derived] Taylor MK, Sullivan DK, Swerdlow RH, Vidoni ED, Morris JK, Mahnken JD, Burns JM. A high-glycemic diet is associated with cerebral amyloid burden in cognitively normal older adults. Am J Clin Nutr. 2017 Dec;106(6):1463-1470. doi: 10.3945/ajcn.117.162263. Epub 2017 Oct 25. PMID 29070566

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise Group | Control Group
Started | 78 | 39
Completed | 75 | 34
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise Group | Control Group | Total
Number analyzed (Participants) | 78 | 39 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 78 | 39 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (5.3) | 71.2 (4.8) | 71.5 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 24 | 79
  Male | 23 | 15 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 78 | 39 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 77 | 35 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 78 | 39 | 117

OUTCOME MEASURES:

1. Primary Outcome: Amyloid Burden
Description: Amyloid burden measure is mean Florbetapir cortical-to-cerebellar uptake ratio averaged across 6 regions of interest (frontal, temporal, parietal, anterior cingulate, posterior cingulate, and precuneus). Higher numbers mean more amyloid accumulation. There is no defined maximum value. Zero is the theoretical minimum value.
Time Frame: Baseline to 52 weeks
Population: Six individuals did not complete follow-up testing due to withdrawal. Two refused follow-up PET.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value Ratio (SUVR)
Arm/Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 74 | 35
Standard Uptake Value Ratio (SUVR)
  Baseline | 1.20 (.2) | 1.22 (.2)
  Follow-up | 1.21 (.2) | 1.22 (.2)

2. Secondary Outcome: Whole Brain Volume
Description: Whole brain volume in mL define by Freesurfer analysis. Higher numbers indicate greater brain volume. There is no defined maximum. Zero is the theoretical minimum.
Time Frame: Baseline to 52 weeks
Population: Six individuals did not complete follow-up testing due to withdrawal. Seven refused follow-up MRI.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 70 | 34
mL
  Baseline | 1068.7 (109.7) | 1061.7 (114.4)
  Follow-up | 1063.4 (109.1) | 1059.1 (115.1)

3. Secondary Outcome: Executive Function
Description: Executive Function ability to be measured using confirmatory factor analysis (CFA). CFA aggregates scores from across multiple subtests. Values are standard deviations centered on a pooled baseline (all participant scores at baseline). Higher values mean improvement over baseline testing. Lower scores (including negative) mean worse performance after baseline testing. There is no minimum or maximum score.
Time Frame: Baseline to Week 52
Population: Six individuals did not complete follow-up testing due to withdrawal.
Measure: Mean (Standard Deviation); unit: Standard Deviations
Arm/Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 75 | 36
Standard Deviations
  Baseline | 0.029 (.46) | -0.042 (.37)
  Week 26 | 0.017 (0.63) | -0.035 (0.39)
  Follow-up | .018 (.62) | -0.037 (0.45)

ADVERSE EVENTS:
Time Frame: One year
Description: Adverse events were defined and graded according to CTCAE 3.0
Arm/Group | Aerobic Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/39
Serious Adverse Events (participants affected / at risk) | 8/78 | 4/39
Other Adverse Events (participants affected / at risk) | 23/78 | 4/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise Group (N=78) | Control Group (N=39)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Grade 3 Supraventricular Tachycardia
Infection with unknown ANC (Infections and infestations) | 4 (4) | 1 (1) — Grade 3 Post-surgical infection with unknown
Lower extremity arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Grade 3 lower extremity arthroplasty (1 knee, 1 hop
Hepatobiliary inflammation (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 3Ibuprofen toxicity and liver inflammation
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Grade 3 Breast Cancer
Acute Pyelonephritis with urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Grade 3Acute Pyelonephritis with urinary tract infection
Fall and hip fracture requiring fixation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Fall and hip fracture requiring fixation Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise Group (N=78) | Control Group (N=39)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (23) | 4 (4) — Joint pain - Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT02000583/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT02000583/Prot_SAP_001.pdf